CLINICAL TRIAL: NCT01168284
Title: A Coping Effectiveness Training Intervention for Caregivers of Children With Autism Spectrum Disorders: A Feasibility Study
Brief Title: A Coping Effectiveness Training Intervention for Caregivers of Children With Autism Spectrum: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Purpose: Other
Other Study IDs: 999910160; 10-HG-N160
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-11-21

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

INTERVENTIONS:
Behavioral: Coping Effectiveness Training

SUMMARY:
In recent years, there have been a growing number of individuals diagnosed with Autism Spectrum Disorders (ASD). As such, this increase has expanded the number of caregivers of children with ASD. Research has shown that having a child with an ASD is stressful for caregivers and their families. More specifically, prior research suggests that caregivers of children with ASD may find it difficult to maintain feelings of control and to cope with the overall physical and emotional demands of caring for their child. A previous study of caregivers of children with ASD found that caregivers felt a lack of personal control over aspects of their child s condition and also found it difficult to cope with various demands of caregiving. Furthermore, this study found that greater levels of perceived personal control and the use of problem-focused coping strategies were associated with caregivers adaptation to their child s condition. As such, the goal of our research is to conduct a feasibility study using a coping effectiveness training (CET) intervention designed to enhance perceived personal control (PPC) and coping efficacy in caregivers of children with ASD. There has been a growing interest in developing interventions targeted at constructs involved in the adaptation process. However, there have been few studies of interventions targeting predictors of adaptation such as PPC and coping efficacy. Research has shown that the CET intervention can enhance coping efficacy in several other populations. This intervention also incorporates appraisals of one s ability to change a particular situation. The conceptual framework for our study was adapted from Lazarus and Folkman s Transactional Model of Stress and Coping. A cross-sectional randomized treatment-control design is proposed to evaluate the use of a CET intervention intended to enhance PPC and coping efficacy. Caregivers of children with ASD will be recruited from support groups, autism resource centers, and four clinics. Participants randomized to the treatment group will be asked to complete baseline and follow-up surveys and two 1.5-hour individualized in-person sessions. Participants randomized to the control group will be asked to complete baseline and follow-up surveys and two 1.5-hour individualized in-person client-centered discussion sessions. The main outcome measures will be participation, reasons for withdrawal, participants experiences within the intervention setting and their experiences in applying the intervention, PPC, coping efficacy, and coping effectiveness.

DETAILED DESCRIPTION:
In recent years, there have been a growing number of individuals diagnosed with Autism Spectrum Disorders (ASD). As such, this increase has expanded the number of caregivers of children with ASD. Research has shown that having a child with an ASD is stressful for caregivers and their families. More specifically, prior research suggests that caregivers of children with ASD may find it difficult to maintain feelings of control and to cope with the overall physical and emotional demands of caring for their child. A previous study of caregivers of children with ASD found that caregivers felt a lack of personal control over aspects of their child s condition and also found it difficult to cope with various demands of caregiving. Furthermore, this study found that greater levels of perceived personal control and the use of problem-focused coping strategies were associated with caregivers adaptation to their child s condition. As such, the goal of our research is to conduct a feasibility study using a coping effectiveness training (CET) intervention designed to enhance perceived personal control (PPC) and coping efficacy in caregivers of children with ASD. There has been a growing interest in developing interventions targeted at constructs involved in the adaptation process. However, there have been few studies of interventions targeting predictors of adaptation such as PPC and coping efficacy. Research has shown that the CET intervention can enhance coping efficacy in several other populations. This intervention also incorporates appraisals of one s ability to change a particular situation. The conceptual framework for our study was adapted from Lazarus and Folkman s Transactional Model of Stress and Coping. A cross-sectional randomized treatment-control design is proposed to evaluate the use of a CET intervention intended to enhance PPC and coping efficacy. Caregivers of children with ASD will be recruited from support groups, autism resource centers, and four clinics. Participants randomized to the treatment group will be asked to complete baseline and follow-up surveys and two 1.5-hour individualized in-person sessions. Participants randomized to the control group will be asked to complete baseline and follow-up surveys and two 1.5-hour individualized in-person client-centered discussion sessions. The main outcome measures will be participation, reasons for withdrawal, participants experiences within the intervention setting and their experiences in applying the intervention, PPC, coping efficacy, and coping effectiveness.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must be a primary caregiver (biological or adoptive parent or grandparent) of a child with an ASD [note: no restrictions with regard to age of the child or how recently s/he was diagnosed
* Must be at least 18 years of age
* Caregivers must reside with the child
* Only one caregiver per household and this person should be the caregiver that spends the most time with the child.
* Must be able to read, write, and speak English

EXCLUSION CRITERIA:

- Those who have a child with any specific genetic diagnosis associated with ASD [including Rett, Tuberous Sclerosis Complex, Fragile X Syndrome, Neurofibromatosis, Prader-Willi Syndrome, and Angelman Syndrome will not be eligible to participate in this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-07-05; Primary Completion 2011-04-04 (Actual); Study Completion 2011-05-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Astin JA, Beckner W, Soeken K, Hochberg MC, Berman B. Psychological interventions for rheumatoid arthritis: a meta-analysis of randomized controlled trials. Arthritis Rheum. 2002 Jun 15;47(3):291-302. doi: 10.1002/art.10416. PMID 12115160
- [Background] Chesney MA, Neilands TB, Chambers DB, Taylor JM, Folkman S. A validity and reliability study of the coping self-efficacy scale. Br J Health Psychol. 2006 Sep;11(Pt 3):421-37. doi: 10.1348/135910705X53155. PMID 16870053
- [Background] Hall S, Reid E, Ukoumunne OC, Weinman J, Marteau TM. Brief smoking cessation advice from practice nurses during routine cervical smear tests appointments: a cluster randomised controlled trial assessing feasibility, acceptability and potential effectiveness. Br J Cancer. 2007 Apr 10;96(7):1057-61. doi: 10.1038/sj.bjc.6603684. PMID 17406348